CLINICAL TRIAL: NCT02178969
Title: A Prospective Short-term Study to Evaluate Methodologies for the Assessment of Disease Extent, Impact, and Wound Evolution in Patients With Dystrophic Epidermolysis Bullosa (DEB)
Brief Title: Short Term Observational Study in DEB Patients
Status: Completed | Type: Observational
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Other Study IDs: SHP-608-002
Record Dates: First submitted 2014-06-04; First posted 2014-07-01 (Estimated); Last update posted 2021-03-17 (Actual); Status verified 2021-03

CONDITIONS: Dystrophic Epidermolysis Bullosa
MeSH Terms: conditions — Epidermolysis Bullosa Dystrophica

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Optional genetic test for DEB diagnosis
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to better understand disease extent and to identify appropriate methodologies to evaluate (dystrophic epidermolysis bullosa) DEB in a quantitative and qualitative manner.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent is provided. Patients 18 years of age and older, and parent(s)/legal guardian(s) of patients younger than 18 years of age, must provide written informed consent prior to participating in the study; additionally, informed assent will be obtained from patients younger than 18 years of age as specified by local requirements.
2. Patient must have a documented diagnosis of DEB based on genetic analysis showing a mutation in COL7A1 or, in the opinion of the investigator, a confirmed diagnosis of DEB based on histologic criteria (antigen mapping or electron microscopy).
3. Patient must have at least 5 wounds that are suitable for imaging, in the opinion of the investigator, at the time of enrollment.
4. Patient is willing and able to undergo the protocol-specified procedures.

Exclusion Criteria:

1. Patient has used or is currently using experimental treatment for DEB including, but not limited to, bone marrow transplantation, systemic immune suppression, or experimental procedures that involve live cells, with potential for systemic spread such as gene transfer, stem cell infusions, or other cell type injections such that, in the opinion of the investigator, inclusion poses an unacceptable risk to the patient or interpretation of these study data.
2. Patient has squamous cell carcinoma with evidence of locally invasive disease or distant metastases.
3. Patient is pregnant.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with DEB.
Sampling Method: Non-Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2014-06-24 (Actual); Primary Completion 2015-02-23 (Actual); Study Completion 2015-02-23 (Actual)

PRIMARY OUTCOMES:
Wound Surface Area (WSA) of patient- and investigator-selected wounds | Over 4 weeks
Wound Surface Area (WSA) as a percentage of Body Surface Area (BSA) in patients with DEB | Over 4 weeks

SECONDARY OUTCOMES:
The number, severity and relationship to study procedures of adverse events (AEs) and serious AEs (SAEs) | Over 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (10):
- United States (3):
  - Ann and Robert H Lurie Childrens Hospital of Chicago, Chicago, Illinois
  - Columbia University Medical Center, New York, New York
  - Cincinnati Childrens Hospital Medical Center, Cincinnati, Ohio
- Premier Specialists Pty Ltd, Kogarah, Australia
- Salzburger Landeskliniken, Salzburg, Austria
- Fakultni nemocnice Brno, Brno, Czechia
- Service de Génétique et INSERM UMR 1163, Laboratoire de Génétique des maladies cutanées - Institut Imagine, Paris, France
- Universitätsklinikum Freiburg, Freiburg im Breisgau, Germany
- Italy (2):
  - Ospedale Pediatrico Bambino Gesù, Roma
  - Istituto Dermopatico Dell'immacolata IRCCS, Rome

REFERENCES:
- [Derived] Paller AS, Pope E, Rudin D, Malyala A, Ramsdell D, Johnson R, Landy H, Murrell DF; DEB Investigators. A prospective short-term study to evaluate methodologies for the assessment of disease extent, impact, and wound evolution in patients with dystrophic epidermolysis bullosa. Orphanet J Rare Dis. 2022 Aug 13;17(1):314. doi: 10.1186/s13023-022-02461-z. PMID 35964087
- See also: To obtain more information on the study, click here/on this link. — https://clinicaltrials.takeda.com/study-detail/5f6b5fd54db2bf003ab46de2